CLINICAL TRIAL: NCT00465517
Title: A Double-blind, Randomized, Placebo-controlled Study to Evaluate the Safety, Tolerability, and Efficacy of Ganaxolone as add-on Therapy in Adult Subjects With Epilepsy Consisting of Uncontrolled Partial-onset Seizures.
Brief Title: A Randomized, Controlled Trial of Ganaxolone in Adult Uncontrolled Partial-Onset Seizures
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Marinus Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1042-0600; V 1.3
Record Dates: First submitted 2007-04-24; First posted 2007-04-25 (Estimated); Results first posted 2023-03-15 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-02

CONDITIONS: Partial Epilepsy; Catamenial Epilepsy
Keywords: Partial onset seizures; Complex-partial seizures; Anticonvulsant; Partial seizures; Catamenial epilepsy
MeSH Terms: conditions — Epilepsies, Partial; Seizures | interventions — ganaxolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ganaxolone (Experimental): active study drug
  Interventions: Drug: Ganaxolone
- non-active drug (Placebo Comparator): placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Ganaxolone — Oral suspension 200-500 mg 3x/day
  Arms: ganaxolone
Other: Placebo — non-active placebo
  Arms: non-active drug

SUMMARY:
The study will evaluate the effectiveness and safety of an investigational drug-ganaxolone - on partial seizure frequency in adults with epilepsy taking a maximum of 3 antiepileptic medications (AEDs). The study will also evaluate the effectiveness of ganaxolone in females with catamenial epilepsy.

Catamenial epilepsy refers to a relationship between seizure frequency and a woman's menstrual cycle, where the number of seizures increases around the time of a woman's menstrual cycle.

ELIGIBILITY:
INCLUSION CRITERIA:

* Diagnosis of epilepsy with POS with or without secondary generalized seizures according to the International League Against Epilepsy [ILAE] Classification of Epileptic Seizures (1981). Diagnosis should have been established by clinical history and CT or MRI of the brain to rule out progressive structural lesions and EEG with results consistent with partial-onset epilepsy.
* During the 8 week baseline period preceding randomization visit (Visit 4), participants should have a documented seizure frequency of ≥ 3CPS per 4 weeks on average.
* Participants should not be seizure free for more than 28 consecutive days during treatment with a stable dose of AEDs [Note: Participants with historically sufficiently high seizure frequency who fall short 1 seizure in any 4 weeks period or with a seizure-free period > 28 consecutive days may be allowed to enter the study after discussion with the Medical Monitor. Prolongation of the screening period for questionable cases may also be allowed by the Medical Monitor.]
* Treatment with a stable dose of up to 3 (FDA approved) current AEDs for 1 month prior to screening.
* Maintenance of current AEDs without a change in dosing for the duration of study.

  * Concomitant vigabatrin not permitted;
  * Felbamate is allowed if the participant has been on felbamate for at least 18 months and has stable laboratory tests) for the course of the study. [Note: A shorter period for stable laboratory results may be allowed by the Medical Monitor, depending on the extent of dose change and the half-life of the AED.]
  * Participants receiving treatment with a vagal nerve stimulator (VNS) may be included as long as the VNS has been in place for at least 12 months prior to entry into the study, the VNS battery is not due for replacement during 0600 subject participation, and stimulation parameters have been kept constant for 1 month prior to screening. VNS will be counted as 1 of the 3 concomitant AEDs.
* Male or female, 18 to 69 years of age (inclusive). [Note: Participants who are > 69 years of age but are of good health condition may be allowed to enter the study after discussion with and approval by the Medical Monitor.]
* A 12-lead electrocardiogram (ECG) w/o clinically significant abnormalities.
* Be properly informed of the nature and risks of the study and give informed consent in writing, prior to entering the study.
* Able to participate for the full term of study.
* Able to keep a seizure & medication diary throughout the course of the study.
* Sexually active women of childbearing potential (WCBP) must be using a medically acceptable method of birth control and have a negative qualitative β-human chorionic growth hormone (β-HCG) pregnancy test result from a urine sample collected at the initial screening visit. A woman of childbearing potential is defined as a female who is biologically capable of becoming pregnant. A medically acceptable method of birth control includes intrauterine devices in place for at least 3 months, surgical sterilization, or adequate barrier methods (e.g., diaphragm and foam). An oral contraceptive alone is not considered adequate for the purpose of this study. Use of oral contraceptives in combination with another method (eg, a spermicidal cream) is acceptable.in participants who are not sexually active, abstinence is an acceptable form of birth control and serum β-HCG must be tested per protocol.
* Participants with a history of depression who are stable and may be taking 1 anti-depressant medication.

EXCLUSION CRITERIA:

* Presence of non-motor simple partial seizures only.
* History of pseudoseizures in the last 5 years.
* History of a primary generalized seizure in the last 5 years.
* Past use of vigabatrin without stable visual fields tested twice over the 12 months after the last dose of vigabatrin (Concomitant use of vigabatrin is not allowed).
* Seizures secondary to illicit drug or alcohol use, infection, neoplasia, demyelinating disease, degenerative neurological disease, or CNS disease deemed progressive, metabolic illness, or progressive degenerative disease.
* Status epilepticus within the last year prior to randomization.
* Clinically unstable psychiatric disorder within the last 2 years.
* Suicidal attempt within the last 5 years or current significant suicidal ideation.
* History of psychosis within the last 5 years. [Note: Participants who suffered a psychosis that can well be explained by exogenous factors may be allowed to enter the study after discussion with and approval by the Medical Monitor.]
* Current use of neuroleptics for psychosis.
* A significant medical or surgical condition at screening which might compromise the hematologic, cardiovascular, pulmonary, renal, gastrointestinal, or hepatic systems or other conditions that would place the subject at increased risk.
* Known sensitivity or allergy to progesterone or related steroid compounds.
* History of drug use or alcohol abuse within the past 5 years.
* Sexually active WCBP who are unwilling to use a double-barrier method and establish that they are currently not pregnant by submitting to a pregnancy test.
* Females who are currently breastfeeding.
* history of chronic noncompliance with drug regimens.
* Exposure to any other investigational drug or device within 30 days prior to screening.
* Alanine transferase (ALT; SGPT) or Aspartate transferase (AST; SGOT) levels > 3 times upper limits of normal (ULN) at screening.
* Benzodiazepines may be used intermittently for the control of seizure clustering as a one time rescue up to a maximum of 4 occasions as follows:

  * Participants who need benzodiazepines for control of seizures more than once per month or more than 4 times total during the Titration and Maintenance Phases will be discontinued.
  * Once during the Titration Phase
  * No more than once per month during the Maintenance Phase
  * Each occasion may be a period of 24 hours, during which up to 3 doses of benzodiazepine may be used.
  * If a participant is taking a benzodiazepine chronically for epilepsy and non-epilepsy conditions, it will be counted as 1 of the 3 AEDs and the dose cannot be changed during the study.
* Participant has history of repetitive seizures within the 12-month period preceding study entry where the individual seizures cannot be counted.
* Inability to withhold grapefruit and grapefruit juice from diet for the entire clinical trial.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2007-02; Primary Completion 2008-10 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (27):
- United States (27):
  - University of Alabama, Birmingham, Alabama
  - Barrow Neurological Institute, Phoenix, Arizona
  - Arkansas Epilepsy Program, Little Rock, Arkansas
  - University of Southern California Adult Comprehensive Epilepsy Center, Los Angeles, California
  - University of California-Davis, Sacramento, California
  - Anchutz Outpatient Pavillion Neurosciences Clinic/ University of Colorado Hospital, Aurora, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - University of Florida McKnight Brain Institute, Gainesville, Florida
  - Intercoastal Medicine, Sarasota, Florida
  - Emory HealthCare, Atlanta, Georgia
  - Southern Illinois University Medical Center, Springfield, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kentucky, Dept. of Neurology, Lexington, Kentucky
  - Mid-Atlantic Epilepsy and Sleep Center, Bethesda, Maryland
  - 2799 West Grand blvd. CFP 071, Detroit, Michigan
  - Minnesota Epilepsy Group, PA, Saint Paul, Minnesota
  - Comprehensive Epilepsy Care Center for Children and Adults, Chesterfield, Missouri
  - Overlook Hospital and Hackensack Medical Center, Hackensack, New Jersey
  - Neurosciences Institute at Albany Medical Center, Albany, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Ohio State University Medical Center, Columbus, Ohio
  - Riddle Health Care Center for Neuroscience, Media, Pennsylvania
  - Drexel University / Hahneman Hospital, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Ctr, Nashville, Tennessee
  - Neurological Clinic of Texas, P.A., Dallas, Texas
  - Virginia Commonwealth University, Richmond, Virginia

REFERENCES:
- [Derived] Maguire MJ, Nevitt SJ. Treatments for seizures in catamenial (menstrual-related) epilepsy. Cochrane Database Syst Rev. 2021 Sep 16;9(9):CD013225. doi: 10.1002/14651858.CD013225.pub3. PMID 34528245
- See also: information about ganaxolone — https://marinuspharma.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: No recruitment details specified
Pre-assignment Details: Participants were randomized (Visit 4, Week 0, before dosing) to receive investigational product in an active:placebo ratio of 2:1.
Groups:
- Ganaxolone: Suspension formulation 50 milligrams per milliliter (mg/mL) three times daily (TID)
- Placebo: Placebo Suspension 50 mg/mL TID
Period: Overall Study
Arm/Group | Ganaxolone | Placebo
Started | 98 | 49
Completed | 86 | 45
Not Completed | 12 | 4
Not completed — Adverse Event | 7 | 3
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 4 | 1

BASELINE CHARACTERISTICS:
Population: ITT Population: All randomized participants who received at least 1 dose of study medication.
Groups:
- Ganaxolone: Suspension formulation 50 mg/mL TID
- Total: Total of all reporting groups
Arm/Group | Ganaxolone | Placebo | Total
Number analyzed (Participants) | 98 | 49 | 147
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.1 (11.74) | 40.2 (11.11) | 39.5 (11.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 36 | 100
  Male | 34 | 13 | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 4 | 11
  Not Hispanic or Latino | 91 | 45 | 136
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 4 | 12
  White | 87 | 42 | 129
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 3 | 5
Region of Enrollment [Number; unit: participants]
  United States | 98 | 49 | 147

OUTCOME MEASURES:

1. Primary Outcome: Mean Weekly Log-transformed Seizure Frequency During Weeks 1 Through 10
Description: Weekly seizure frequency, analyzed as mean weekly log-transformed seizure frequency [including partial-onset seizures (POS) with or without secondary generalization, but not non-motor simple partial seizure (SPS)] during Weeks 1 through 10.
Time Frame: Week 1 through Week 10
Population: ITT Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: log[seizures per week]
Arm/Group | Ganaxolone | Placebo
Number analyzed (Participants) | 98 | 48
log[seizures per week] | 5.20 (9.286) | 10.77 (44.156)

2. Secondary Outcome: Mean Weekly Log-transformed Seizure Frequency During Weeks 3 Through 10
Description: Weekly seizure frequency, analyzed as mean weekly log-transformed seizure frequency [including POS with or without secondary generalization, but not non-motor SPS] during the Weeks 3 through 10
Time Frame: Week 3 through Week 10
Population: Only those participants with data available during Weeks 3 to 10 were analyzed.
Measure: Mean (Standard Deviation); unit: log[seizures per week]
Arm/Group | Ganaxolone | Placebo
Number analyzed (Participants) | 95 | 46
log[seizures per week] | 5.44 (9.431) | 11.90 (50.209)

3. Secondary Outcome: Change From Baseline in Mean Weekly Seizure Frequency During Weeks 1 Through 10
Description: Summary of change from Baseline in mean weekly seizure frequency is presented. Baseline was defined as the Day 0 assessment before study drug infusion. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline and at Week 1 through Week 10
Population: ITT Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Seizures per week
Arm/Group | Ganaxolone | Placebo
Number analyzed (Participants) | 98 | 48
Seizures per week | -1.27 (3.567) | 1.41 (15.075)

4. Secondary Outcome: Change From Baseline in Mean Weekly Seizure Frequency During Weeks 3 Through 10
Description: as for outcome 3
Time Frame: Baseline and at Week 3 through Week 10
Population: Only those participants with data available during Weeks 3 to 10 were analyzed.
Measure: Mean (Standard Deviation); unit: Seizures per week
Arm/Group | Ganaxolone | Placebo
Number analyzed (Participants) | 95 | 46
Seizures per week | -1.07 (3.909) | 2.52 (20.229)

5. Secondary Outcome: Percent Change From Baseline in Mean Weekly Seizure Frequency During Weeks 1 Through 10
Description: Summary of percent change from Baseline in mean weekly seizure frequency is presented. Baseline was defined as the Day 0 assessment before study drug infusion. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline and at Week 1 through Week 10
Population: ITT Population. Only those participants with data available at the specified data points were analyzed
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Ganaxolone | Placebo
Number analyzed (Participants) | 98 | 48
Percent change | -17.59 (48.867) | 1.99 (63.160)

6. Secondary Outcome: Percent Change From Baseline in Mean Weekly Seizure Frequency During Weeks 3 Through 10
Description: as for outcome 5
Time Frame: Baseline and at Week 3 through Week 10
Population: Only those participants with data available during Weeks 3 to 10 were analyzed.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Ganaxolone | Placebo
Number analyzed (Participants) | 95 | 46
Percent change | -12.08 (54.286) | 4.57 (71.880)

7. Secondary Outcome: Mean Weekly Seizure Frequency for Each Week After Dosing During Weeks 1 to 10
Description: Mean weekly Seizure Frequency for each week post-dosing During Weeks 1 to 10 is presented.
Time Frame: Weeks 1, 2, 3, 4, 5, 6, 7, 8, 9 and 10
Population: ITT Population. Only those participants with data available at the specified data points were analyzed
Measure: Mean (Standard Deviation); unit: Seizures per week
Arm/Group | Ganaxolone | Placebo
Number analyzed (Participants) | 98 | 48
Seizures per week
  Week 1: number analyzed (Participants) | 96 | 48
  Week 1 | 4.53 (11.195) | 7.25 (21.668)
  Week 2 | 5.09 (9.638) | 8.79 (34.548)
  Week 3: number analyzed (Participants) | 95 | 46
  Week 3 | 5.02 (9.743) | 7.80 (28.163)
  Week 4: number analyzed (Participants) | 95 | 45
  Week 4 | 5.69 (10.738) | 9.13 (30.768)
  Week 5: number analyzed (Participants) | 93 | 45
  Week 5 | 5.12 (9.085) | 11.64 (42.864)
  Week 6: number analyzed (Participants) | 91 | 45
  Week 6 | 5.65 (8.894) | 10.43 (38.133)
  Week 7: number analyzed (Participants) | 91 | 45
  Week 7 | 6.68 (10.894) | 13.15 (62.762)
  Week 8: number analyzed (Participants) | 87 | 45
  Week 8 | 4.63 (8.401) | 13.47 (63.157)
  Week 9: number analyzed (Participants) | 87 | 45
  Week 9 | 5.07 (9.897) | 11.64 (49.387)
  Week 10: number analyzed (Participants) | 85 | 44
  Week 10 | 4.83 (9.282) | 13.60 (56.711)

8. Secondary Outcome: Percent Change From Baseline in Mean Weekly Seizure Frequency by Subtype During Weeks 1 Through 10
Description: Seizure subtypes included Complex partial seizures (CPS), Generalized tonic-clonic seizure (GTCS), and Simple partial seizure (SPS)-motor. Percent Change from Baseline in Mean Weekly Seizure frequency by seizure subtype is presented. Baseline was defined as the Day 0 assessment before study drug infusion. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline and at Week 1 through Week 10
Population: Only those participants with data available during Weeks 1 to 10 were analyzed.
Measure: Mean (Standard Error); unit: Percent change
Arm/Group | Ganaxolone | Placebo
Number analyzed (Participants) | 96 | 47
Percent change
  CPS | -17.47 (51.055) | 3.88 (82.986)
  GTC: number analyzed (Participants) | 23 | 14
  GTC | -30.65 (79.104) | -37.75 (64.091)
  SPS-motor: number analyzed (Participants) | 37 | 21
  SPS-motor | -30.63 (81.214) | 19.70 (195.966)

9. Secondary Outcome: Number of Responders During Weeks 1 Through 10
Description: Responders were defined as participants experiencing ≥50% of reduction in mean weekly seizure frequency from the Baseline. Baseline was defined as the Day 0 assessment before study drug infusion.
Time Frame: Baseline and at Week 1 through Week 10
Population: ITT Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Ganaxolone | Placebo
Number analyzed (Participants) | 98 | 49
Participants | 23 | 7

10. Secondary Outcome: Number of Responders During Weeks 3 Through 10
Description: as for outcome 9
Time Frame: Baseline and at Week 3 through Week 10
Population: ITT Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Ganaxolone | Placebo
Number analyzed (Participants) | 98 | 49
Participants | 25 | 6

11. Secondary Outcome: Number of Seizure-free Participants Up to Week 2
Description: Number of seizure-free participants is presented.
Time Frame: Up to Week 2
Population: Only those participants with data available Up to week 2 were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Ganaxolone | Placebo
Number analyzed (Participants) | 95 | 48
Participants | 16 | 4

12. Secondary Outcome: Number of Seizure-free Participants During Weeks 3 Through 10
Description: Number of seizure-free participants is presented.
Time Frame: Week 3 through Week 10
Population: Only those participants with data available during Weeks 3 to 10 were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Ganaxolone | Placebo
Number analyzed (Participants) | 95 | 46
Participants | 0 | 1

13. Secondary Outcome: Number of Seizure-free Participants During Weeks 1 Through 10
Description: Number of seizure-free participants is presented.
Time Frame: Week 1 through Week 10
Population: ITT Population. Only those participants with data available at the specified data points were analyzed
Measure: Count of Participants; unit: Participants
Arm/Group | Ganaxolone | Placebo
Number analyzed (Participants) | 98 | 48
Participants | 1 | 0

14. Secondary Outcome: Number of Seizure-free Days Up to Week 2
Description: Summary of Seizure-Free days is presented.
Time Frame: Up to Week 2
Population: Only those participants with data available up to Week 2 were analyzed.
Measure: Mean (Standard Deviation); unit: Seizure free days
Arm/Group | Ganaxolone | Placebo
Number analyzed (Participants) | 95 | 48
Seizure free days | 10.3 (4.41) | 10.0 (3.78)

15. Secondary Outcome: Number of Seizure-free Days During Week 3 Through 10
Description: Summary of Seizure-Free days is presented.
Time Frame: Week 3 through Week 10
Population: Only those participants with data available during Weeks 3 to 10 were analyzed.
Measure: Mean (Standard Deviation); unit: Seizure free days
Arm/Group | Ganaxolone | Placebo
Number analyzed (Participants) | 95 | 46
Seizure free days | 37.1 (18.50) | 38.5 (16.17)

16. Secondary Outcome: Number of Seizure-free Days During Week 1 Through 10
Description: Summary of Seizure-Free days is presented.
Time Frame: Week 1 through Week 10
Population: ITT Population. Only those participants with data available at the specified data points were analyzed
Measure: Mean (Standard Deviation); unit: Seizure free days
Arm/Group | Ganaxolone | Placebo
Number analyzed (Participants) | 98 | 48
Seizure free days | 45.9 (22.11) | 46.8 (20.59)

ADVERSE EVENTS:
Time Frame: Screening through Week 14
Description: Adverse events (AEs) and Serious adverse events (SAEs) were collected for ITT Population which consisted of all randomized participants who received at least 1 dose of study medication.
Arm/Group | Ganaxolone | Placebo
All-Cause Mortality (participants affected / at risk) | 0/98 | 0/49
Serious Adverse Events (participants affected / at risk) | 5/98 | 4/49
Other Adverse Events (participants affected / at risk) | 82/98 | 38/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ganaxolone (N=98) | Placebo (N=49)
Brain contusion (Injury, poisoning and procedural complications) | 1 | 0
Burns second degree (Injury, poisoning and procedural complications) | 0 | 1
Hemothorax (Injury, poisoning and procedural complications) | 1 | 0
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 1 | 0
Subdural hematoma (Injury, poisoning and procedural complications) | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Enteritis (Gastrointestinal disorders) | 0 | 1
Epilepsy (Nervous system disorders) | 1 | 0
Migraine (Nervous system disorders) | 0 | 1
Postictal state (Nervous system disorders) | 1 | 0
Hematocrit decreased (Investigations) | 1 | 0
Hemaglobin decreased (Gastrointestinal disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Mediastinal shift (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary hematoma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ganaxolone (N=98) | Placebo (N=49)
Dizziness (Nervous system disorders) | 16 | 4
Headache (Nervous system disorders) | 8 | 6
Somnolence (Nervous system disorders) | 13 | 1
Convulsion (Nervous system disorders) | 5 | 4
Coordinate abnormal (Nervous system disorders) | 6 | 3
Nystagmus (Nervous system disorders) | 3 | 3
Sedation (Nervous system disorders) | 4 | 0
Balance disorder (Nervous system disorders) | 3 | 0
Tremor (Nervous system disorders) | 2 | 1
Amnesia (Nervous system disorders) | 2 | 0
Dysarthria (Nervous system disorders) | 2 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 1
Memory Impairment (Nervous system disorders) | 2 | 0
Aphasia (Nervous system disorders) | 1 | 0
Cervicogenic headache (Nervous system disorders) | 0 | 1
Cognitive disorder (Nervous system disorders) | 1 | 0
Complex partial seizures (Nervous system disorders) | 0 | 1
Grand mal convulsion (Nervous system disorders) | 0 | 1
Intention tremor (Nervous system disorders) | 0 | 1
Lethargy (Nervous system disorders) | 1 | 0
Mental impairment (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 1
Postictal headache (Nervous system disorders) | 0 | 1
Sinus headache (Nervous system disorders) | 1 | 0
Fatigue (General disorders) | 16 | 4
Irritability (General disorders) | 4 | 1
Adverse drug reaction (General disorders) | 3 | 1
Pyrexia (General disorders) | 2 | 1
Feeling drunk (General disorders) | 2 | 0
Gait disturbance (General disorders) | 0 | 2
Chest pain (General disorders) | 0 | 1
Feeling cold (General disorders) | 1 | 0
Influenza like illness (General disorders) | 1 | 0
Local swelling (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Pain (General disorders) | 1 | 0
Pitting oedema (General disorders) | 1 | 1
Tenderness (General disorders) | 0 | 1
Flatulence (Gastrointestinal disorders) | 3 | 3
Nausea (Gastrointestinal disorders) | 4 | 2
Constipation (Gastrointestinal disorders) | 2 | 3
Abdominal pain upper (Gastrointestinal disorders) | 2 | 2
Diarrhoea (Gastrointestinal disorders) | 3 | 0
Stomach discomfort (Gastrointestinal disorders) | 1 | 2
Abdominal distension (Gastrointestinal disorders) | 1 | 1
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0
Abdominal tenderness (Gastrointestinal disorders) | 0 | 1
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 1
Dry mouth (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Faeces discoloured (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Lip disorder (Gastrointestinal disorders) | 0 | 1
Lip swelling (Gastrointestinal disorders) | 1 | 0
Oral pain (Gastrointestinal disorders) | 1 | 0
Paraesthesia oral (Gastrointestinal disorders) | 1 | 0
Submaxillary gland enlargement (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 1
Nasopharyngitis (Infections and infestations) | 5 | 5
Sinusitis (Infections and infestations) | 2 | 3
Upper respiratory tract infection (Infections and infestations) | 2 | 3
Influenza (Infections and infestations) | 1 | 2
Gastroenteritis viral (Infections and infestations) | 1 | 1
Urinary tract infection (Infections and infestations) | 1 | 1
Gastroenteritis (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0
Infected insect bite (Infections and infestations) | 1 | 0
Kidney infection (Infections and infestations) | 0 | 1
Postoperative wound infection (Infections and infestations) | 1 | 0
Rhinitis (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 1 | 0
Tooth infection (Infections and infestations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 5 | 6
Skin laceration (Injury, poisoning and procedural complications) | 5 | 0
Contusion (Injury, poisoning and procedural complications) | 2 | 1
Skeletal injury (Injury, poisoning and procedural complications) | 1 | 1
Animal bite (Injury, poisoning and procedural complications) | 1 | 0
Ear abrasion (Injury, poisoning and procedural complications) | 1 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 1
Face injury (Injury, poisoning and procedural complications) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 1
Joint sprain (Injury, poisoning and procedural complications) | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0
Sunburn (Injury, poisoning and procedural complications) | 0 | 1
Depression (Psychiatric disorders) | 4 | 0
Insomnia (Psychiatric disorders) | 0 | 3
Abnormal dreams (Psychiatric disorders) | 1 | 1
Affective disorder (Psychiatric disorders) | 1 | 1
Confusional state (Psychiatric disorders) | 2 | 0
Affect liability (Psychiatric disorders) | 0 | 1
Aggression (Psychiatric disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 1 | 0
Dysphemia (Psychiatric disorders) | 0 | 1
Libido decreased (Psychiatric disorders) | 1 | 0
Mental state changes (Psychiatric disorders) | 1 | 0
Mood altered (Psychiatric disorders) | 1 | 0
Stress (Psychiatric disorders) | 1 | 0
Tearfulness (Psychiatric disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 1
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Hypotrichosis (Skin and subcutaneous tissue disorders) | 1 | 0
Increased tendency to bruise (Skin and subcutaneous tissue disorders) | 1 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Vision blurred (Eye disorders) | 5 | 0
Diplopia (Eye disorders) | 3 | 1
Eye swelling (Eye disorders) | 1 | 0
Oscillopsia (Eye disorders) | 1 | 0
Visual disturbance (Eye disorders) | 1 | 0
Ammonia increased (Investigations) | 1 | 0
Blood glucose abnormal (Investigations) | 1 | 0
Weight increased (Investigations) | 1 | 0
White blood cell count decreased (Investigations) | 1 | 0
Genital pruritus female (Reproductive system and breast disorders) | 2 | 0
Breast tenderness (Reproductive system and breast disorders) | 1 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 0
Menstrual disorder (Reproductive system and breast disorders) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 2 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Dysuria (Metabolism and nutrition disorders) | 1 | 1
Nephrolithiasis (Metabolism and nutrition disorders) | 1 | 0
Hypertension (Vascular disorders) | 2 | 0
Hot flush (Vascular disorders) | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 1
Dysmorphism (Congenital, familial and genetic disorders) | 0 | 1
Goitre (Endocrine disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Multiple allergies (Immune system disorders) | 0 | 1
Tooth extraction (Surgical and medical procedures) | 0 | 1

LIMITATIONS AND CAVEATS:
Overall count of AEs provided is associated with 'at least 1 AE'.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less